CLINICAL TRIAL: NCT01486316
Title: Integrated Diagnostic Evaluation in Non-Therapy DevIces For the studY of Heart Failure
Brief Title: Diagnostic Device Risk Management of Atrial Fibrillation and Heart Failure
Acronym: IDENTIFY-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IDENTIFY-HF
Record Dates: First submitted 2011-11-04; First posted 2011-12-06 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Atrial Fibrillation; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Other): Subjects in the Control arm will be observed between implant and month 12. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location). At month 12 through study close (month 18), study doctors for the all subjects will have access to the risk status.
  Interventions: Device: Reveal XT® Insertable Cardiac Monitor; Other: Heart Failure Risk Status Diagnostic
- Risk Status Guided (Experimental): Study doctors will have access to the experimental IDENTIFY-HF Risk Status for subjects in the Guided arm between months 6 and 18. At all times during the study, study doctors will also be able to use the standard device diagnostics in the office using the programmer, or by data transmission from the patient's home (or another remote location).
  Interventions: Device: Reveal XT® Insertable Cardiac Monitor; Other: Heart Failure Risk Status Diagnostic

INTERVENTIONS:
Device: Reveal XT® Insertable Cardiac Monitor — If not previously implanted, a non-experimental insertable cardiac monitor will be implanted to collect information on the patients' heart condition as inputs into the heart failure risk status algorithm (during guided follow-up only, Guided arm: 6-18 months, Control arm: 12-18 months).
  Other Names: Reveal XT®
Other: Heart Failure Risk Status Diagnostic — The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status and standard device trend data are provided to study doctors for remote management of their patients' heart failure using study specific protocols. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".

SUMMARY:
The purpose of this study is to characterize the feasibility and impact of a diagnostic tool that may help clinicians identify when patients are at higher risk of visiting the hospital for a heart failure event. The study will use a non-experimental device that is inserted just under the skin of the chest, which continuously monitors the heart rhythm in combination with an experimental web-based heart failure risk status. Patients with atrial fibrillation and heart failure will be evaluated to collect data about the potential of this risk status to help improve patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient (or patient's legally authorized representative) is willing and able to provide written informed consent
* Patient is willing and able to comply with the protocol, including follow-up visits
* Documented paroxysmal or persistent atrial fibrillation or strong suspicion of atrial fibrillation (i.e, palpitations)
* Patient is indicated for the Reveal XT insertable cardiac monitor or other commercially-available and substantially equivalent Medtronic insertable cardiac monitor
* Recent HF event within prior 120 days (HF event defined as meeting any one of the following two criteria: 1. Admission with primary diagnosis of HF 2. Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any one of the following settings: admission with secondary/tertiary diagnosis of HF, emergency department, ambulance, observation unit, urgent care, HF/cardiology clinic, patient's home
* Willing and able to transmit data via CareLink

Exclusion Criteria:

* Patient is pregnant
* Patient has been participating in another study that may interfere with the IDENTIFY-HF protocol required procedures
* Endstage (Stage D or New York Heart Association class IV) heart failure
* Asymptomatic (Stage B or New York Heart Association class I) heart failure
* Severe aortic stenosis or insufficiency
* Existing insertable cardiac monitor implanted for more than 1 year
* Existing implantable pulse generator, implantable cardioverter defibrillator, cardiac resynchronization therapy device
* Severe renal impairment (estimated glomerular filtration rate <25mL/min)
* Myocardial infarction within prior 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: IDENTIFY-HF Team, Study Chair — Medtronic
Locations (11):
- United States (11):
  - Scripps Green, La Jolla, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Spectrum Health, Grand Rapids, Michigan
  - The Valley Hospital, Ridgewood, New Jersey
  - Carolinas Medical Center/Sanger Heart & Vascular, Charlotte, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Lancaster Heart & Stroke Foundation, Lancaster, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Thomas Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Heart Clinic PLLC, McAllen, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: The Control arm will be observed between implant and month 12. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location). At month 12 through study close (month 18), study doctors for the all subjects will have access to the risk status.
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
- Risk Status Guided: Study doctors will have access to the experimental IDENTIFY-HF Risk Status for subjects in the Guided arm between months 6 and 18. At all times during the study, study doctors will also be able to use the standard device diagnostics in the office using the programmer, or by data transmission from the patient's home (or another remote location).
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
- No Implant: Subjects who did not undergo an implant attempt and were not randomized.
- Implanted Not Randomized: Subject were implanted and not randomized
Period: Overall Study
Arm/Group | Control Arm | Risk Status Guided | No Implant | Implanted Not Randomized
Started | 7 (prior to study closure, 24 subjects were enrolled 7 subjects randomized to Control Arm) | 10 (prior to study closure, 24 subjects were enrolled with 10 being randomized to HFRS Guided Arm) | 5 (Exited prior to implant) | 2 (Exited prior to 6 month visit)
Completed (18 Month/Exit Visit) | 3 | 7 | 0 | 0
Not Completed | 4 | 3 | 5 | 2
Not completed — Device explanted with/without re-implant | 3 | 2 | 0 | 2
Not completed — Not meeting eligibility criteria | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Arm: Subjects in the Control arm will be observed between implant and month 12. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location). At month 12 through study close (month 18), study doctors for the all subjects will have access to the risk status.
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
- Not Randomized: Subjects who were not randomized
- Total: Total of all reporting groups
Arm/Group | Control Arm | Risk Status Guided | Not Randomized | Total
Number analyzed (Participants) | 7 | 10 | 7 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (7.6) | 66.2 (15.3) | 70.3 (9.7) | 69.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 3 | 6 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 10 | 7 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
New York Heart Assocation (NYHA) Functional Classification [Number; unit: number] — NYHA Class is a measure of a patient's degree of heart failure with 4 possible scores, ranging from I to IV. The classifications and 2015 definitions are as follows:
  I: No limitation of physical activity. II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest.
  number
    NYHA Class II | 5 | 6 | 3 | 14
    NYHA Class III | 2 | 4 | 4 | 10
LVEF [Mean (Standard Deviation); unit: percentage] | 60.0 (4.1) | 60.2 (10.7) | 50.6 (11.6) | 57.3 (10.2)
Heart Failure Stage [Number; unit: Participants]
  Stage C | 6 | 9 | 5 | 20
  Not available | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Heart Failure Risk Score (HFRS) With Heart Failure Events
Description: Evaluate the HFRS Algorithm prior to Heart Failure (HF) related clinical events among patients with HF and documented or suspected AF. Daily HFRS scores were calculated each day for each patient with an implanted Reveal XT device, and the scores were ordinal, with possible values of "Low", "Medium", "High", and "Very High". The objective was to assess the association between the daily scores before and after HF events (HF-related hospitalizations, clinic visits) among subjects experiencing such visits. This would only be done during follow-up periods in which physicians were blinded to the scores (see Time Frame). The score could only be generated if the subject performed a CareLink transmission of their device data during follow-up.
  Because of the small number of subjects enrolled, formal statistical analyses were not performed. Subjects were partitioned by whether they (1) experienced a HF event, and (2) whether they experienced a High or Very High HFRS score.
Time Frame: 0 to 6 months post-implant (HFRS Guided Arm), 0-12 months (Control Arm)
Measure: Number; unit: participants
Groups:
- Control Arm: The Control arm will be observed between months 13-18. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location), but study doctors for the subjects will have access to the risk status.
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
Arm/Group | Control Arm | Risk Status Guided
Number analyzed (Participants) | 7 | 10
participants
  High/Very High Score & HF Event(s) | 5 | 2
  High/Very High Score, No HF Event(s) | 2 | 7
  HF Event(s), No High/Very High Score | 0 | 0
  No High/Very High Score or HF Event(s) | 0 | 1

2. Other Pre Specified Outcome: Correlation of HFRS Status With Actions/Testing
Description: At scheduled visits in which the HFRS scores were available to clinicians, the scores were summarized, along with whether subjects experienced significant weight gain, high blood pressure, or reported heart failure symptoms.
  Because of the small number of subjects randomized, no formal statistical analyses were performed.
Time Frame: 6 to 18 months post-implant (HFRS Guided Arm), 13-18 months (Control Arm)
Population: Only randomized subjects who did not exit prior to the period in which clinicians could utilized the HFRS score (6-18 months for HFRS Guided Arm, 13-18 months for Control Arm) were included in the analysis.
Measure: Number; unit: Visits with high/very high score
Units Other Than Participants: Visits with High/Very High HFRS Score
Groups:
- Control Arm: The Control arm will be observed between months 13-18, and so only the subjects followed beyond 12 months are included in the analysis. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location), but study doctors for the subjects will have access to the risk status.
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
Arm/Group | Control Arm | Risk Status Guided
Number analyzed (Participants) | 4 | 10
Number analyzed (Visits with High/Very High HFRS Score) | 3 | 58
Visits with high/very high score
  Significant Weight Gain Reported | 0 | 9
  High Blood Pressure | 0 | 5
  HF Symptoms Reported | 1 | 46
  Medications Adjusted due to HFRS Score | 1 | 18
  Rate Control Meds Adjusted due to HFRS Score | 0 | 1
  Blood Pressure Meds Adjusted due to HFRS Score | 0 | 4
  Diuretics Adjusted due to HFRS Score | 1 | 15
  Directed to Clinic | 0 | 9
  Directed to Emergency Department | 0 | 0
  Directed to Hospital | 0 | 0

3. Other Pre Specified Outcome: Clinical Status Measures
Description: Characterize the difference in clinical status measures over time in each arm. Outcomes include Quality of Life (as measured by the Minnesota Living With Heart Failure Questionnaire, in which scores range from 0 (Best) to 105 (Worst), 6 Minute Hall Walk distance, and New York Heart Association (NYHA, ranging from Class I (Best) to Class IV (Worst))
  Because of the small number of patients enrolled, formal statistical analyses were not performed and data were not summarized in aggregate.
Time Frame: 0 to 18 months post-implant
Population: Subjects randomized to the Risk Status Guided Arm
Measure: Count of Units; unit: Outcome of Patients During Guided Period
Units Other Than Participants: Outcome of Patients During Guided Period
Groups:
- Control Arm: The Control arm will be observed between months 13-18, and so only Control arm subjects followed beyond 12 months are included. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location), but study doctors for the subjects will have access to the risk status.
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status. The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
Arm/Group | Risk Status Guided | Control Arm
Number analyzed (Participants) | 10 | 4
Number analyzed (Outcome of Patients During Guided Period) | 25 | 2
Outcome of Patients During Guided Period
  HF Event During Guided Period | 6 | 1
  High/Very High HFRS Score During Guided Period | 7 | 1
  Quality of Life Improvement During Guided Period | 5 | 0
  6 Minute Hall Walk Improved During Guided Period | 3 | 0
  Improved NYHA During Guided Period | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the point of enrollment to the completion of follow-up (18 months).
Description: All subjects were assessed for adverse events through their follow-up visits as well as unscheduled visits as the adverse events occurred.
Groups:
- Control Arm: Subjects in the Control arm will be observed between implant and month 12. During this time, the standard device diagnostic suite will be used as it would normally, in the office using the programmer, or by data transmission from the patient's home (or another remote location). At month 12 through study close (month 18), study doctors for the all subjects will have access to the risk status.
  Heart Failure Risk Status Diagnostic: The experimental IDENTIFY-HF Risk Status developed for this study will be used to change standard device data to a heart failure risk status.The risk status inputs are: night heart rate, heart rate variability, atrial fibrillation burden, ventricular rate during atrial fibrillation, patient activity.
  Based on pre-defined thresholds for each of the above inputs, as well as data trends, a heart failure score is derived. The heart failure score is then classified as: "Low", "Medium", "High", or "Very High".
Arm/Group | Control Arm | Risk Status Guided
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 6/7 | 5/10
Other Adverse Events (participants affected / at risk) | 6/7 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=7) | Risk Status Guided (N=10)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Unstable Angina (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fribrillation (Cardiac disorders) | 2 (2) | 2 (3)
Cardiac Failure (Cardiac disorders) | 1 (1) | 4 (4)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
International normalizes ratio decreased (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Vascular Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Endocrine disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=7) | Risk Status Guided (N=10)
Atrial Fribillation (Cardiac disorders) | 4 (6) | 4 (4)
Cardiac Failure (Cardiac disorders) | 3 (7) | 3 (3)
Drug Intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Chest Discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cough (General disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No